CLINICAL TRIAL: NCT07114263
Title: Study of The Analgesic Profile of Two Adjuvants Added to Low Dose Hyperbaric Bupivacaine Versus One Adjuvant in Patients Undergoing Anal Surgery Using Spinal Anesthesia ( Saddle Block ): A Randomized Prospective Study
Brief Title: Study of The Analgesic Profile of Two Adjuvants Added to Low Dose Hyperbaric Bupivacaine Versus One Adjuvant in Patients Undergoing Anal Surgery Using Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ezzat Nasr Ezzat Alhelw, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36264MS785/12/24
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Spinal Anesthesia Administration; Analgesic; Anorectal Surgery
Keywords: anorectal surgeries.; hyperbaric bupivacaine; Dexmedetomidine; Spinal Anesthesia; Saddle Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, anesthesia administrator, and outcome assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group F :Fentanyl group (Experimental): Patients will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5% and 0.5 ml (25 mcg) Fentanyl and 1 ml glucose 5% with total volume of 3ml.
  Interventions: Drug: Group F (fentanyl group)
- Group D: Dexmedetomidine group (Experimental): Patients will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5% and 1 ml (4 mcg) Dexmedetomidine and 0.5 ml glucose 5% with total volume of 3ml.
  Interventions: Drug: Group D :Dexmedetomidine group
- Group DF :Fentanyl and Dexmedetomidine (Experimental): Patients will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5%, 0.5 ml (25 mcg) Fentanyl and 1 ml (4 mcg) Dexmedetomidine with total volume of 3ml.
  Interventions: Drug: Group DF :Fentanyl and Dexmedetomidine group

INTERVENTIONS:
Drug: Group F (fentanyl group) — Group F (fentanyl group):will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5% and 0.5 ml (25 mcg) Fentanyl and 1 ml glucose 5% with total volume of 3ml.
  Arms: Group F :Fentanyl group
Drug: Group D :Dexmedetomidine group — Group D :Dexmedetomidine group: will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5% and 1 ml (4 mcg) Dexmedetomidine and 0.5 ml glucose 5% with total volume of 3ml.
  Arms: Group D: Dexmedetomidine group
Drug: Group DF :Fentanyl and Dexmedetomidine group — Fentanyl and Dexmedetomidine group:will receive intrathecal 1.5 ml hyperbaric bupivacaine 0.5%, 0.5 ml (25 mcg) Fentanyl and 1 ml (4 mcg) Dexmedetomidine with total volume of 3ml.
  Arms: Group DF :Fentanyl and Dexmedetomidine

SUMMARY:
This study will be conducted to compare the efficacy of fentanyl and Dexmedetomidine as an additive to hyperbaric bupivacaine 0.5% in saddle block anesthesia on duration of analgesia in patients undergoing anorectal surgeries.

DETAILED DESCRIPTION:
Pilonidal sinus, hemorrhoidectomy, anal fistula or fissure repair are the main types of anorectal surgery. Various surgical and anesthetic techniques have been introduced to improve analgesia level and limit the motor blockade.Regional anesthesia is preferred for anorectal surgeries to avoid the risks of general anesthesia. Besides, providing effective post-operative analgesia, regional techniques reduce the opioid use.

Intrathecal administration of drugs to obtain anesthesia has been in use since the turn of the twelfth century. Saddle block anesthesia is a kind of low spinal block that provides anesthesia over the saddle area, i.e., perineum, perianal area, medial aspect of legs and thigh.

Saddle block anesthesia is performed by injecting a small dose of hyperbaric local anaesthetic at the level of L3, L4 after which the patient is maintained in sitting position for a few minutes to facilitate preferential impregnation of sacred roots (S1 to S5), which is responsible for innervation of perineum, external genitalia and anus. The saddle block causes a parasympathetic blockade at the bladder level which may result in bladder and rectal atony which is advantageous because of sphincteric relaxation needed for the operation.

Hyperbaric bupivacaine 0.5% is the most common local anaesthetic used for spinal anaesthesia for lower abdominal and lower limb surgeries. One disadvantage with using hyperbaric bupivacaine alone is a relatively shorter duration of action that means that early analgesic intervention is needed in postoperative period. Adjuvants are drugs that increase the efficacy or potency of other drugs when given concurrently. Neuraxial adjuvants are used to increase the speed of the onset of neural blockade (reduce latency), improve the quality and prolong the duration of neural blockade.

Fentanyl is a lipophilic short-acting opioid that exhibits close structural similarities to local anesthesia and has demonstrable local anesthetic efficacy on sensory C primary afferent nerve fibers, which may facilitate analgesic effects. It has improved spinal anesthesia and reduced the anesthetic drug related side effects including pruritus, nausea and vomiting.

Dexmedetomidine, a highly selective alpha_2 agonist, is being introduced as an adjuvant to local anesthetics with significant analgesic, sympatholytic, and sedative properties. Compared to clonidine; Dexmedetomidine is approximately eight times more selective towards α2-adrenergic receptors , which is associated with sedative and analgesic effects in supraspinal and spinal sites and also has an antinociceptive impact on both visceral and somatic pain.

This study will be conducted to compare the efficacy of fentanyl and Dexmedetomidine as an additive to hyperbaric bupivacaine 0.5% in saddle block anesthesia on duration of analgesia in patients undergoing anorectal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* aged from 18 to 65 years
* American Society of Anesthesiologists' physical I or II of both sexes
* Patients who will be scheduled to surgery for their uncomplicated hemorrhoids, anal fissure, or anal fistula in lithotomy position will be included in the study.

Exclusion Criteria:

* Infection focus at back, history of spine surgery, coagulopathy, mental disturbance, and neurological disease.
* drug allergy.
* intake of experimental or analgesic medication within last 24 hours.
* patients receiving alpha-adrenergic antagonist will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 2 hours
  from time of spinal block to first demand of rescue analgesia

SECONDARY OUTCOMES:
Incidence of complications | 24 hours
  c) Incidence of complications e.g., Hypotension, Bradycardia, nausea/vomiting, urinary retention, pruritus, and shivering.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF